CLINICAL TRIAL: NCT06724510
Title: Safety and Efficacy Evaluation of High Intensity Focused Ultrasound Device in Eyebrow Lifting, a Prospective, Multi-center, Evaluator Blinded, Randomized, Non-treatment Controlled, and Superiority Clinical Trial
Brief Title: Safety and Efficacy Evaluation of High Intensity Focused Ultrasound Device in Eyebrow Lifting
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: CLASSYS Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CLSGQDWJJCHS
Record Dates: First submitted 2024-12-01; First posted 2024-12-09 (Actual); Last update posted 2025-04-25 (Actual); Status verified 2025-03

CONDITIONS: Skin Laxity; Wrinkles; Facial Wrinkles and Rhytides Reduction
Keywords: High Intensity Focused Ultrasound; HIFU; ULTRAFORMER MPT; ULTRAFORMER; MPT; Eyebrow; Eyebrow Lifting
MeSH Terms: conditions — Cutis Laxa

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- ULTRAFOMER MPT (Experimental): This arm receives the high-intensity focused ultrasound (HIFU) treatment, which is the primary intervention being evaluated for efficacy and safety in eyebrow lifting.
  Interventions: Device: HIFU treatment with ULTRAFOMER MPT
- No Treatment (No Intervention): This arm does not receive any treatment, serving as a comparison group to evaluate the efficacy of the investigational device.

INTERVENTIONS:
Device: HIFU treatment with ULTRAFOMER MPT — The high-intensity focused ultrasound (HIFU) treatment, which is the primary intervention being evaluated for efficacy and safety in eyebrow lifting.
  Arms: ULTRAFOMER MPT

SUMMARY:
The goal of this clinical trial is to assess the safety and efficacy of the high-intensity focused ultrasound (HIFU) device, ULTRAFORMER MPT (UF4-M400), developed by CLASSYS Inc., for eyebrow lifting. This study is a prospective, multicenter, evaluator-blinded, randomized, non-treatment-controlled, superiority clinical trial.

The main questions the study seeks to answer are:

Does the ULTRAFORMER MPT device effectively lift eyebrows? Is the safety profile of the ULTRAFORMER MPT device acceptable? Researchers will compare the investigational device to a non-treatment control group to determine whether the HIFU device demonstrates superiority in eyebrow lifting outcomes.

Participant Details:

Participants will receive a single treatment session using the investigational device or be assigned to the non-treatment control group.

Follow-up will occur over 3 months to evaluate the effectiveness and safety of the treatment.

Outcomes:

Primary Outcome: Eyebrow lifting improvement, assessed through standardized photographic evaluation and other aesthetic measurement tools.

Secondary Outcomes: Participant satisfaction using the Global Aesthetic Improvement Scale (GAIS) and pain assessment using a Visual Analog Scale (VAS).

Safety Measures: Monitoring for adverse events (AEs) and serious adverse events (SAEs) throughout the study period.

This trial aims to provide robust evidence supporting the use of the ULTRAFORMER MPT for non-invasive eyebrow lifting.

ELIGIBILITY:
Inclusion Criteria:

1. Age: 20 to 65 years old at the time of consent.
2. Condition: Forehead skin laxity with Forehead Lines Grading Scale score of 1-3.
3. Consent: Ability to understand trial details, voluntarily participate, and comply with treatment and follow-up.

Exclusion Criteria:

1. Skin Conditions: Hyperpigmentation, tattoos, scars, active skin diseases, or other conditions (e.g., eczema, psoriasis, vitiligo) in the treatment area that may affect efficacy or increase risk.
2. Medical Devices or Implants: Presence of metal implants or embedded electronic devices in the treatment area.
3. Health Conditions: Severe dysfunction of vital organs (e.g., heart, liver, kidneys), autoimmune diseases, or uncontrolled diabetes.
4. Medications: Recent use of anti-thrombotic agents, NSAIDs, or other drugs affecting coagulation within one week before screening.
5. Prior Treatments: Use of fillers (e.g., hyaluronic acid, collagen) or cosmetic procedures (e.g., laser therapy, botulinum toxin) in the treatment area within the specified timeframes.
6. Pregnancy: Women who are pregnant, nursing, or not using birth control during the trial.

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2024-11-18 (Actual); Primary Completion 2025-04-30 (Estimated); Study Completion 2025-10-31 (Estimated)

PRIMARY OUTCOMES:
Global Aestetic Improvement Scale(GAIS) | 3 months after treatment
  Improvement was defined as GAIS score≤3 Min 1 Max 5
  1. Very much improved
  2. Much improved
  3. Improved
  4. No Change
  5. Worse

CONTACTS AND LOCATIONS:
Overall Officials: Wenzhi Li, Study Chair — Beijing Anzhen Hospital
Locations (3):
- China (3):
  - Beijing Anzhen Hospital of Capital Medical University, Beijing
  - TheThird Hospital of Hebei Medical University, Shijiazhuang
  - The Second Affiliated Hospital of Xian Jiaotong University, Xi'an